

Title: A Prospective, Multicenter, Observational Study in Relapsed and/or Refractory Multiple Myeloma Patients Treated with Ixazomib plus Lenalidomide and Dexamethasone

NCT Number: NCT03433001

Statistical analysis plan Approve Date: 01-NOV-2021

Certain information within this statistical analysis plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).

Note; This document was translated into English as the language on original version was Japanese.

# to the applicable Terms of Use my L: A Prospective, Multicenter, Observational Study in Relapsed and/or Refractory Multiple Myeloma Patients Treated with Ixazomib plus Lenalidomide and Dexamethasone

(Study number: C16042)

# Statistical Analysis Plan

(Ver.3.0; NOV 01, 2021)

Secondary Sponsor: Takeda Pharmaceutical Company Limited

Property of Takeda. For non-commercial use only and subject to the

| | TEDMS and Abbrevia | tions | 1 |
|---|---|---|---|
| | Analysis sets | RAPHICS AND OTHER BASELINE ents tion Patients Patients | 4 |
| 4 | Considerations for ano | Avoic | 4 |
| · | other data handling | 11ySIS | 4 |
| _ | DATIENTS DEMOC | DADILICS AND OTHER DASELINE | 5 |
| | PATIENTS, DEMOG | RAPHICS AND OTHER BASELINE | 14 0 |
| • | HAKACIEKISIICS | | A C |
| | 5.1 Disposition of Pati | ents | .01 |
| | 5.1.1 Study Informa | ition | 11 |
| | 5.1.2 Eligibility of F | ratients | 11 |
| | 5.1.3 Exit Status of | Patients | 11 |
| | 5.1.4 Protocol Devia | ations and Analysis Datasets | 12 |
| | 5.2.1 Demographics | and Other Baseline Characteristics | 13 |
| | 5.2.2 Cytogenetic A | bnormalities | 14 |
| | 5.2.3 Comorbidity | | 14 |
| | 5.2.4 Prior Therapy. | | 15 |
| | 5.2.5 Supportive Th | erapy | 16 |
| | 5.2.6 Next-line Trea | atment | 16 |
| ( | Eficacy Analysis | bnormalities | 17 |
| | 6.1 Primary Endpoint | and Analytical Methods | 17 |
| | 6.2 Supplemental Anal | lysis for Primary Endpoint | 17 |
| | 6.3 Secondary Endpoin | nts and Analytical Methods | 17 |
| | 6.3.1 PFS rate at 12 | and 24 Months from the Start of Study Treatment | 17 |
| | 6.3.2 Subgroup anal | ysis of PFS from the Start of Study Treatment | 18 |
| | 6.3.3 OS from the S | tart of Study Treatment | 18 |
| | 6.3.4 Best Response | <u>, </u> | 19 |
| | 6.3.5 Time to Next | Treatment (TTNT) | 19 |
| | 6.3.6 Duration of Th | herapy (DOT) | 20 |
| | 6.3.7 Proportion of 1 | Patients Continuing Treatment at 12 and 24 Months from | the |
| | Start of Study Treatme | ent | 20 |
| | 629 Oyumall Dagma | nse Rate (ORR) | |
| | 6.3.9 Very Good Pa | rtial Response (VGPR) or More | 21 |
| | 6.3.10 Patient Report | ted Outcome Health-related Quality of Life (HRQol): | |
| , 0 | EORTC-QLQ-C30/M | Y-20 | 21 |
| KY, | 6.3.11 Proportion of 1 | Patients with CR who Achieve Minimal Residual Disease | |
| Property | (MRD) Negativity in I | Bone Marrow | |
| 0101 | 6.3.12 Relative Dose | Intensity (RDI) | |
| X | 6.3.13 Imaging Evalu | ation | |
| | 1 | | |

| 6.3 | 3.15 Duration of Response (DOR) | | 23 |
|---|---|---|---|
| 6.3 | 3.16 Examination of Prognostic Factors Rega | arding PFS, OS, TTNT and | DOR24 |
| 7 Sa | ıfety analysis | | 25 |
| 7.1 | Frequency of Treatment-Emergent Adverse | Event | 25 |
| 7.1 | 1.1 Overview of Treatment-Emergent Adve | erse Event | 25 |
| 7.1 | 1.2 Output of Treatment-Emergent Adverse | Event | 25 |
| 7.2 | Laboratory Results | | 26 C |
| 8 Li | stings | | 27 |
| 9 Co | onsiderations on Statistical Analysis | | 27 |
| 9.1 | Covariate | i,C | 27 |
| 9.2 | Handling of Dropouts or Missing Data | | 27 |
| 9.3 | Criteria for Interim Analysis and Early Disc | ontinuation | 27 |
| 9.4 | Multicenter Studies | 1/0 | 27 |
| 9.5 | Multiple Comparisons/Multiplicity | XO | 27 |
| 9.6 | Consideration of Subgroups | | 27 |
| 10 Re | evision history | | 27 |
| Property | 3.16 Examination of Prognostic Factors Registery analysis | | |

# 1 TERMS AND ABBREVIATIONS

Summary Statistics: number, mean, standard deviation, minimum/maximum value, quartiles

Full Analysis Set (FAS): All patients who enroll into the study and who receive at least one dose of ixazomib. Patients with enrollment violation will be excluded.

Evaluable Analysis Set: All patients included in the FAS who have mean start of IRd therapy and who have at least one Safety Analysis Set: Safety Analysis Set: All patients who enroll into the study who receive at least one dose of any drug used in IRd therapy (i.e. ixazomib, lenalidomide, or dexamethasone).

# 3 CONSIDERATIONS FOR ANALYSIS

Significance level

5% (one-sided test)

Confidence coefficient

For only primary analysis, 90% (two-sided estimation)

Otherwise, 95% (two-sided estimation)

Number of display digits

The significant digit is the lowest digit included in each variable of data unless otherwise specified; if the values "160" and "160.1" are included, the first decimal place will be the significant digit.

Mean/Quartiles/Confidence interval Round off two digits below the effective digit of the data and display up to one digit below.

Standard deviation

Round off the third digit below the effective digit of the data and display up to the second digit below.

Minimum/Maximum value

Display up to the significant digit of data.

Proportion/Percentage

Round off the second decimal place and display to the first decimal place.

P value

Round off the 5 decimal places and display up to 4 decimal places. However, when p value is less than 0.0001, it represents as "p < 0.0001."

# 4 OTHER DATA HANDLING

- Duration
- Duration (day)

Target Date - Start Date + 1

- > TEAE
- TEAE (treatment-emergent adverse event)
   AE that occurred from the start of IRd treatment until 30 days after the end of IRd treatment or the start of next treatment, whichever occurs first.
- Relative dose intensity (RDI)
- RDI

$$RDI(\%) = \frac{\text{(Actual dose)/(Actual number of cycle days)}}{\text{(Scheduled dose)/(Scheduled number of cycle days)}} \times 100$$

The actual number of cycle days shall be (next cycle start date) - (relevant cycle start date) if there is a next course, or the number of scheduled cycle days if there is no next course. The number of scheduled cycle days and dose for each drug should be set as following table.

| | Drug | Length of cycle | Dose |
|-----|---------------|-----------------|---------|
| | Ixazomib | | 4.0mg×3 |
| IRd | Lenalidomide | 28 | 25mg×21 |
| | Dexamethasone | | 40mg×4 |

# > Frailty

The score of frailty should be set as following table. As a sensitivity analysis, changes in age categories may be considered.

| categories in | ay be considered. | | |
|---------------------|-------------------|-------------|-------|
| 4 | Ite | ems | Score |
| , Å· | | 75<= | 0 |
| Property of Lakeda. | Age | 76<= - <=80 | 1 |
| | | <=81 | 2 |
| | ADL | 4<= | 1 |
| | | <=5 | 0 |
| | IADL | 5<= | 1 |
| | | <=6 | 0 |
| RIC | CCI | 1<= | 0 |
| ▼ | | <=2 | 1 |
| The 4.4.1 | | | |

The total score will be classified as follows.

Properly of Takeda: For non-confinercial use only and subject to the applicable Terms of Use

# Cytogenetic risk

Expanded high risk group
Patients with abnormalities in either one of del17p, t(4;14), t(14;16) or 1q gain Modified Standard risk group
All other patients

Renal function
ation for the exti Patients are classified into High risk group and Standard risk group, or Expanded high risk group and Modified Standard risk group according to the pattern of chromosome aberrations at the time of recurrence.

- High risk group
- Expanded high risk group
- Modified Standard risk group

# 

Calculation for the estimation of eGFR, published by the Japanese Society of Nephrology (2008):

For men:

eGFR (mL/min/1.73 m<sup>2</sup>) = 194 \* serum creatinine [mg/dL]<sup>-1.094</sup> \* age [years]  $^{-0.287}$ 

For Women:

eGFR (mL/min/1.73 m<sup>2</sup>) = 194 \* serum creatinine [mg/dL]<sup>-1.094</sup> \* age [years]<sup>-0.287</sup>×0.739

Cockcroft-Gault equation for the estimation of Ccr:

For men:

Ccr= ((140-age [years])×weight [kg])/(72×serum creatinine [mg/dL])

For women:

((140-age [years])×weight [kg])/(72×serum creatinine [mg/dL])×0.85 Ccr=

Property of Lakeda. Fi Renal function will be classified according to baseline CCr as following table.

| CCr |
|----------|
| 90≦ |
| 60≦ < 90 |
| 30≦ < 60 |
| < 30 |

- Handling of values below or above the quantitative limit
- Serum free light chain (FLC)

If FLC  $\kappa$  or FLC  $\lambda$  is below the limit of quantification, the limit of quantification is imputed.  $\kappa/\lambda$ ratio is calculated using the imputed value.

- International Staging System (ISS)
- Staging criteria (according to Study Protocol Appendix C)

Stage I: (Serum β2-microglobulin <3.5 mg/L) and (Serum albumin ≥3.5 g/dL)

Stage II: Neither Stage I or Stage III

Stage III: Serum β2-microglobulin ≥5.5 mg/L

- I rotocol Appendix C)

  Stage I or Stage III

  There are two definitions of Stage II:

  (serum β2-microglobulin <3.5 mg/dL) and (serum albumin <3.5 g/dL), or serum β2-microglobulin 3.5 -<5.5 mg/dL (irrespective of serum albumin concentrated stage (ISS) at the recurrence (at the start of treatment)

  values. If the patient does not fall into Stage TT albumin is missing, the patient of \* The clinical stage (ISS) at the recurrence (at the start of treatment) is calculated from the clinical laboratory values. If the patient does not fall into Stage III and any one of serum β2-microglobulin and serum albumin is missing, the patient should not be classified.
- Censoring scheme
- Overall survival (OS)

| m albumin is missing, the patient should not be classified. | | |
|---|---|---|
| Censoring scheme verall survival (OS) | | |
| Situation | Date of event expression or censoring | Outcome |
| Death | Date of death | event |
| Discontinuation | Date of discontinuation | - |
| Next antitumor treatment started* | Date of start of next treatment | censoring / - |
| Alive | Last confirmed date of survival | censoring |

For the start coensoring. For the start of next antitumor treatment, analyze both the case of not censoring and the case of

# Progression Free survival (PFS)

| Situation | Date of event expression or censoring | Outcome |
|---|---|---|
| Incomplete or no baseline assessments | Date of first treatment | censoring |
| Progression | Assessment date | event |
| Death | Date of death | event |
| Discontinuation | Date of discontinuation | - |
| Next antitumor treatment started | Date of start of next treatment | censoring |
| No progression | Last confirmed date at which patients are progression-free | censoring |

# Time to Next Treatment (TTNT)

| | | + (/ <sub>1</sub> | |
|---|---|---|---|
| | Situation | Date of event expression or | Outcome |
| | | censoring | |
| | Incomplete or no baseline assessments | Date of first treatment | censoring |
| | Progression | Assessment date | - |
| | Death | Date of death | event |
| | Next antitumor treatment started | Date of start of next treatment | event |
| | Continued study treatment | Last observed date | censoring |
| | Discontinued and no information of next treatment | Last observed date | censoring |
| Last obs | erved date; last date of the date of disconti | nuation, the date of last dose of | study treatment or |
| the date | of final assessment | | |
| Last obsettly of take of | a. Foi no | | |

# Duration of Response (DOR)

DOR is defined for the patients assessed as ≥PR (including patients where two consecutive assessments have not been made) according to the IMWG criteria (2014 version)

| Situation | Date of event expression or | Outcome |
|---|---|---|
| | censoring | |
| Incomplete or no baseline assessments | - | NA 🗸 |
| Progression | Assessment date | event |
| Death | Date of death | event |
| Discontinuation | Date of discontinuation | - 1100 |
| Next antitumor treatment started | Date of start of next | censoring |
| | treatment | 0.1 |
| No progression | Last confirmed date as not | censoring |
| | less than PR | |

# Handling of response assessment

Follow the Research Protocol, Appendix F, Response Criteria [IMWG Criteria (2014 version)]. However, in consideration of the actual clinical situation, the results of only one assessment also will be used for the evaluation that originally "Two consecutive assessments are needed".

- Other valuables to be derived
- Body surface area (BSA)

Property of Takeda. For non-commerce Body Surface Area (m<sup>2</sup>) = Weight (kg)  $^{0.425}$  × Height (cm)  $^{0.725}$  × 0.007184

# 5 PATIENTS, DEMOGRAPHICS AND OTHER BASELINE CHARACTERISTICS

# 5.1 **Disposition of Patients**

# **Study Information** 5.1.1

Analysis Set:

All patients obtained informed consent

Analysis Variables:

The earliest date of informed consent

The latest date of the last visits

Version of MedDRA

Version of SAS

Analysis Methods:

(1) Output above items.

# 5.1.2 **Eligibility of Patients**

Analysis Set:

All patients obtained informed consent

Analysis Variables:

Eligibility [yes, no (reasons)]

Analysis Methods:

(1) Frequency count

# **Exit Status of Patients** 5.1.3

Analysis Set:

Full Analysis Set

Analysis Variables:

Exit status [complete, incomplete (reasons)]

Analysis Methods:

- (1) Frequency count
- (2) Cross table of the number of cycle and the reason for discontinuation

The number of cycles in which any of the drugs of IRd is administered will be used.

Intercial use only and subject to the applicable Terms of Use

# 5.1.4 Protocol Deviations and Analysis Datasets

# **5.1.4.1** Protocol Deviations

Analysis Set:

All patients obtained informed consent

Analysis Variables:

**Protocol Deviations** 

[Major GCP Violations, Deviations of Protocol Entry Criteria, Deviations of Discontinuation Criteria, Deviations Related to Treatment Procedure or Dose, Deviations Concerning Excluded Medication or Therapy, Deviations to Avoid Emergency Risk, Other Deviations]

# Analysis Methods:

(1) Summarize the number of patients who have deviated from the protocol, classify the deviations into above category, and show the breakdown of deviations. Patients applicable for multiple categories will be counted in each category.

# 5.1.4.2 Analysis Datasets

Analysis Set:

All patients obtained informed consent

Analysis Variables:

Protocol deviation related to analysis set [Inclusion, Exclusion]

Inclusion or Exclusion for each analysis set

Full Analysis Set

Evaluable Analysis Set

Safety Analysis Set

Analysis Methods:

Patients applicable for multiple categories will be counted once in each category.

- (1) Frequency count about the determination of inclusion for each analysis set
- (2) Frequency count of the number of patient included for each analysis set

# 5.1.4.3 Patient Flow Diagram

Analysis Set:

All patients obtained informed consent

Analysis Variables:

All patients obtained informed consent

All eligible patients

Age (year) 
$$[Min \le - \le 65, 65 \le - \le 75, 75 \le - \le Max]$$

and Other Baseline Characteristics

...alysis Set, Evaluable Analysis Set, Safety Analysis Set

Analysis Variables:

Age (year) [Min<= -<=65, 65<-<=75, 75<-<=Max]

Sex [Male, Female]

Height (cm)

Veight (kg)

MI (kg/m²)  $^{1}$ 3\(\text{A}(m²)\)

protein isotype [IgG  $\kappa \cdot \lambda$ , IgA  $\kappa_{cl}\lambda$ , IgD  $^{1}$ \(\lambda\$, non-secretory type, unknown) or or all bone marrow plasma cell be mophenotyping: CD20

al stage accor."

il stage.

Clinical stage according to ISS at initial diagnosis [Stage I, II, III]

Clinical stage according to ISS at disease recurrence (at first treatment) [Stage I, II, III]

Chromosome abnormality at the initial diagnosis [t (4;14), t (14;16), t (11;14), del17p, 1q gain]

Chromosomal abnormalities at disease recurrence (at first treatment) [t (4;14), t (14;16), t (11;14),

del17p, 1q gain]

Whether imaging tests are performed [Conducted, Not conducted]

Presence of Bone Lesion [yes, no]

Presence of Extramedullary Masses [yes, no]

Extramedullary Masses [Bone-delivered, Soft tissue-delivered or others]

Prior antineoplastic therapies [Conducted, Not conducted]

Prior radiation therapy [Conducted, Not conducted]

Prior hematopoietic stem cell transplantation [Conducted, Not conducted]

M-protein in blood samples and urine samples

Serum FLC (free light chain) (FLC κ, FLC λ, κ/λ ratio [Min<= - <0.26, 0.26=< - <=1.65, 1.65< - $\leq = Max$ ))

ECOG performance status [0, 1, 2, 3, 4]

Cytogentic risk[High risk, Standard risk], [Expanded high risk, Modified standard risk]

Frequency count of categorical data and summary statistics of continuous data

Note: For patients whose M-protein isotype: type of light chain is "κ", FLC κ will be calculated.

For patients whose M-protein isotype: type of light chain is "λ", FLC λ will be calculated.

Analysis Set:

Full Analysis Set, Evaluable Analysis Set, Safety Analysis Set

Analysis Variables:

Chromosomal abnormalities at disease recurrence (at first treatment) [t/(4;14), t (14;16), t (11;14), del17p, 1q gain]

# Analysis Methods:

- Distribution of chromosomal abnormal cell percentages (1) The distribution of chromosomal abnormal cell percentages is shown in the histogram.
- Frequency count of positive patients of chromosomal abnormalities

The thresholds shall be set as follows,

del17p: 5%

t(4;14), t(14;16), t(11;14), 1q gain: 3%

Frequency count of patterns of chromosomal abnormalities To examine the frequency of combinations of multiple chromosome abnormalities, a frequency count by possible chromosome abnormal pattern will be performed.

# Comorbidity

Analysis Set:

Full Analysis Set

Analysis Variables:

Charlson comorbidity index (CCI);

Myocardial infarction (history, not ECG changes only)

Congestive heart failure

Peripheral disease (includes aortic aneurysm ≥ 6 cm)

Cerebrovascular disease: CVA with mild or no residua or TIA

Dementia

Chronic pulmonary disease

Peptic ulcer disease

.cy. .cy. the applicable Terms of Use applicable Terms of Use applicable Terms of Use applicable Terms of Use Liver disease [Mild (without portal hypertension, includes chronic hepatitis), Moderate or severe]

Diabetes [Without end-organ damage (excludes diet-controlled alone),

With end-organ damage (retinopathy, neuropathy, nephropathy, or brittle diabetes)]

Hemiplegia

Moderate to severe renal disease

Tumor without metastasis (exclude if > 5 years from diagnosis)

Leukemia (acute or chronic)

Lymphoma

Metastatic solid tumor

AIDS (not just HIV positive)

Components of Frailty (Age, ADL, IADL, CCI)

Frailty [Frail, Intermediate fitness, Fit]

# Analysis Methods:

- (1) Frequency count of comorbidity
- Frequency count of components of frailty (2)
- Frequency count[Min<= <=1, - <= Max] and summary statistics of CCI score (3)

# 5.2.4 **Prior Therapy**

Analysis Set:

Full Analysis Set

Analysis Variables:

Prior Antineoplastic Therapies [Bortezomib, Carfilzomib, Lenalidomide, Pomalidomide,

Prednisolone, Dexamethasone, Melphalan, Adriamycin, Cyclophosphamide, Elotuzumab,

Daratumumab, Panobinostat, Vincristine, Other]

Number of collected prior regimen [1, 2, 3, 4.....]

Prior Regimen (Pattern of prior antineoplastic therapies)

Reason for termination by prior regimen (Pattern of prior antineoplastic therapies) [PD or 'other']

Best Response by prior regimen (Pattern of prior antineoplastic therapies) [CR, sCR, ...]

Analysis Methods:

For method (1) and (3), analysis will be performed by one previous drugs, two or more previous regimens and all previous regimens.

Frequency count of prior antineoplastic therapies (1)

<sup>\*</sup>Items with information on severity should be tabulated by severity.

Sorted by frequency. If the antineoplastic therapies is used more than once to the same patient, it will be counted as one case.

3) Summary of prior regimens
For high frequency regimens, the frequency of the regimen, the reason for termination and the response for each regimen will be tabulated.

5.2.5 Supportive Therapy
Analysis Set:
Full Analysis Set

allysis Variables:
upportive Therapy [varicella zoster, P. jirovecii infection (e.g. ST complete)]

allysis Methods:
Frequency regimens will be calculated for each patient, and continued to the calculated.

# Frequency count (1)

Sorted by frequency. If the antineoplastic therapies is used more than once to the same patient, it will be counted as one case.

# Next-line Treatment 3 Set: 5.2.6

Analysis Variables:
Next-line Treat Next-line Treatment [Bortezomib, Carfilzomib, Lenalidomide, Pomalidomide, Prednisolone, Dexamethasone, Melphalan, Adriamycin, Cyclophosphamide, Elotuzumab, Daratumumab, Panobinostat, Vincristine, Other]

Analysis Methods:

# Frequency count

Sorted by frequency. The denominator is the number of patients in the analysis set for which one of the next-line treatments was selected.

# **EFICACY ANALYSIS**

# 6.1 **Primary Endpoint and Analytical Methods**

Analysis Set:

Full Analysis Set

Analysis Variables:

PFS from the start of study Treatment

# Analysis Methods:

icable Terms of Use PFS is defined as the period from the first dose of treatment to the time of confirmed PD or confirmed death (regardless of the cause of death), whichever is earlier. Patients who are still alive and progression-free will be censored at the last confirmed date at which they are progression-free. PFS for the FAS will be estimated using the Kaplan-Meier method, and the quartiles and two-sided 95% confidence intervals will be calculated using the double logarithmic transformation method of Jse only and sulpi Brookmeyer and Crowley.

# **Supplemental Analysis for Primary Endpoint** 6.2

Analysis Set:

Evaluable Analysis Set

Analysis Variables:

PFS from the start of study Treatment

Analysis Methods:

6.1 Analysis will be repeated for Evaluable Analysis Set.

# 6.3 **Secondary Endpoints and Analytical Methods**

# PFS rate at 12 and 24 Months from the Start of Study Treatment

Analysis Set:

Full Analysis Set

Analysis Variables:

PFS rate at Month 12 and 24 from the start of study Treatment

# Analysis Methods:

(1) PFS rate at Month 12, 24 and the two-sided 95% confidence interval will be estimated by Kaplan-Meier method. The confidence interval is constructed based on the variance calculated by Greenwood's formula for the double logarithmically transformed PFS rate, and then calculated by exponential transformation.

# 6.3.2 Subgroup analysis of PFS from the Start of Study Treatment

Analysis Set:

Full Analysis Set, Evaluable Analysis Set

Analysis Variables:

PFS from the start of study Treatment

Strata:

Frailty adjusted group [Fit, Intermediate fitness, Frail]

Cytogenetic risk group [High risk, Standard risk]

Cytogenetic risk group [Expanded High risk, Modified Standard risk]

applicable Terms of Use Chromosomal abnormalities at disease recurrence (at first treatment) [del17p, 1q gain]

Clinical stage according to ISS at disease recurrence (at first treatment) [Stage I, II, III]

Number of regimens [1, 2, 3 or more]

RDI by drug [<80%, >=80%]

Best response [at least VGPR, PR or worse]

Prior antineoplastic therapies\* [Treated, Not treated]

\*Bortezomib, Carfilzomib, Lenalidomide, Pomalidomide, Elotuzumab, Daratumumab

Renal function [Normal, Mild, Moderate, Severe]

Determination of prior treatment efficacy [Clinical relapse, Paraprotein relapse, Other]

# Analysis Methods:

- PFS for each strata will be estimated using similar methodology to that used for analysis of primary analysis. PFS rate at Month 12, 24 and the two-sided 95% confidence interval will be estimated using Kaplan-Meier method.
- Median PFS and the two-sided 95% confidence interval for each strata will be estimated (2) using Brookmeyer and Crowley methodology and display with forest plot.

# 6.3.3 OS from the Start of Study Treatment

Analysis Set:

Full Analysis Set

Analysis Variables:

OS from the start of study Treatment

Analysis Methods:

- (1) OS is defined as the period from the first dose of treatment to the time when death Median OS and the two-sided 95% confidence interval for each strata will be estimated okmeyer and Crowley methodology and display with forest plot.

  est Response
  et:
  sis Sec. 7 (regardless of the cause of death) is confirmed. Patients who are still alive will be censored at the last confirmed date of survival or the date of data cut-off, whichever is earlier. OS for the FAS will be estimated using the Kaplan-Meier method, and the quartiles and two-sided 95% confidence intervals will be calculated using the double logarithmic transformation method of Brookmeyer and Crowley.
- (2)
- and subject to the application and subject to the application of the a (3) using Brookmeyer and Crowley methodology and display with forest plot.

# 6.3.4 **Best Response**

Analysis Set:

Full Analysis Set, Evaluable Analysis Set

Analysis Variables:

Cumulative Best Response

Analysis Methods:

Best response is defined as the cumulative numbers of patients who achieve each level of (1) best response, as defined by the IMWG criteria (2014 version), after each cycle of treatment. A histogram (or similar) showing the numbers of patients achieving different levels of best response will be created after each cycle of treatment.

# Time to Next Treatment (TTNT) 6.3.5

Analysis Set:

Full Analysis Set

Analysis Variables:

Analysis Methods:

TTNT is defined as the period from the first dose of treatment to the time of next-line treatment or confirmed death (regardless of the cause of death), whichever is earlier. Patients who are still alive and no next-line treatment will be censored at the last confirmed date at last observed date. TTNT for the FAS will be estimated using similar methodology to that used for analysis of PFS.

# **Duration of Therapy (DOT)** 6.3.6

Analysis Set:

Full Analysis Set

Analysis Variables:

DOT

# Analysis Methods:

DOT is defined as the treatment duration of IRd therapy. Summary statistics will be (1) calculated. In continuing patients, it is the end of the last cycle with or without drug interrupt. For discontinued patients, the period is defined as the date of IRd initiation to the date of decision to discontinue or the date of the last dose of ixazomib, whichever is later.

# Proportion of Patients Continuing Treatment at 12 and 24 Months from the Start of 6.3.7 and subj **Study Treatment**

Analysis Set:

Full Analysis Set

Analysis Variables:

Proportion of patients continuing treatment with ixazomib at 12 and 24 months from the start of study Treatment

Analysis Methods:

The proportion of patients who are not discontinued at 12 and 24 months after the start of treatment, and the two-sided 95% confidence intervals, will be calculated. Exact confidence intervals will be calculated based on a binomial distribution.

# Overall Response Rate (ORR)

Analysis Set:

Full Analysis Set

Analysis Variables:

# Analysis Methods:

The ORR is defined as the proportion of patients who achieve a best response of PR or better according to the IMWG criteria (2014 version) after the start of the study treatment. The ORR and 95% confidence interval will be calculated. Exact confidence intervals will be calculated based on a binomial distribution.

# 6.3.9 Very Good Partial Response (VGPR) or More

Analysis Set:

Full Analysis Set, Evaluable Analysis Set

Analysis Variables:

Very Good Partial Response (VGPR) or more

# Analysis Methods:

(1) The percentage of patients achieving a VGPR or better, according to the IMWG criteria (2014 version), after the start of the study, and 95% confidence interval will be calculated Exact confidence intervals will be calculated based on a binomial distribution.

# 6.3.10 Patient Reported Outcome Health-related Quality of Life (HRQol): EORTC-QLQ-C30/MY-20

Analysis Set:

Full Analysis Set

Analysis Variables:

EORTC QLQ-C30

- Five functional scales (physical, role, emotional, cognitive, social)
- A global health/quality of life scale
- Three symptom scales (tiredness, nausea and vomiting, pain)
- Six single items (dyspnea, insomnia, anorexia, constipation, diarrhea, economic difficulty)

# **EORTC QLQ-MY20**

- Four independent subscales
- Two functional subscales (body image, future perspective)
- Two symptom subscales (multiple myeloma symptoms, treatment adverse effects)

# Analysis Methods:

- (1) Scores will be calculated for each subscale according to the EORTC Scoring Manual, and summary statistics and 95% confidence intervals will be calculated for each treatment cycle.
- Line plot (Mean  $\pm$  SD) will be presented graphically as plots over time.
- Summary statistics for change from cycle 1, plus the mean and 95% confidence intervals, will be calculated.

# 6.3.11 Proportion of Patients with CR who Achieve Minimal Residual Disease (MRD) Negativity in Bone Marrow

Analysis Set:

Full Analysis Set

Analysis Variables:

Analysis Methods:

The same analysis will be performed for the SRL-flow method and the Adaptive. However, since the quantitative limit of the SRL-flow method is 10<sup>-6</sup>, the smallest category of positive cell rate is tabulated as "less than 10<sup>-6</sup>".

The percentage of corresponding each category will be calculated. 95% confidence (1) interval of percentage of patients achieving MRD negativity will be calculated. Exact confidence intervals will be calculated based on a binomial distribution. If a patient is MRD-positive at their first evaluation and MRD-negative after re-examination, the patient will be considered to be MRDercialuse only and subjection of the contraction of negative and corresponding percentage of MRD positive cells will be used for calculation of the percentage of MRD positive cells

# 6.3.12 Relative Dose Intensity (RDI)

Analysis Set:

Full Analysis Set

Analysis Variables:

**RDI** 

Analysis Methods:

- Summary statistics for RDI for Ixazomib, Lenalidomide and Dexamethasone, will be (1) calculated by cycle.
- Time plot of Analysis (1) will be outputted. (2)
- (3) Summary statistics for RDI for Ixazomib, Lenalidomide and Dexamethasone, will be calculated for overall period.

# 6.3.13 Imaging Evaluation

Analysis Set:

Full Analysis Set

Analysis Variables:

Bone evaluation

**Extramedullary Masses** 

# Analysis Methods:

- , applicable reims of Use The percentage of patients with new bone lesions or extramedullary masses and the twosided 95% confidence intervals will be calculated. Exact confidence intervals will be calculated based on a binomial distribution.
- For the patients with extramedullary masses, frequency count of findings about (2) extramedullary masses will be outputted.

# 6.3.14 M-protein

Analysis Set:

Full Analysis Set

Analysis Variables:

M-protein measurement (SPEP/UPEP [24-hour urine collection], serum free light chain

Best response of SPEP/UPEP percent change

# Analysis Methods:

- Summary statistics and 95% confidence interval of mean will be calculated. (1)
- Summary statistics for change from cycle 1 plus the 95% confidence interval of mean will (2) be calculated.
- The percent change of SPEP/UPEP is achieved when SPEP/UPEP is the lowest value by patients. Summary statistics for percent change from cycle 1 plus the 95% confidence interval of mean will be calculated.

# 6.3.15 Duration of Response (DOR)

Analysis Set:

Full Analysis Set

Analysis Variables:

# Analysis Methods:

DOR is defined as the time from the date of first documentation of response ≥PR according to the IMWG criteria (2014 version) to the date of first documentation of PD or death due to any cause. DOR for patients in the FAS who achieve PR or better at any time during the study will be estimated using the Kaplan-Meier method, and the quartiles and 95% confidence intervals will be calculated by the double logarithmic transformation method of Brookmeyer and Crowley. Patients who achieve PR or better and have not experienced PD will be censored from the date when their response was confirmed as not being worse than PR.

# 6.3.16 Examination of Prognostic Factors Regarding PFS, OS, TTNT and DOR

Analysis Set:

Full Analysis Set

Analysis Variables:

PFS, OS, TTNT and DOR

# Analysis Methods:

cable Terms of Use If necessary, regression analysis using the Cox proportional hazards model will be performed as an exploratory analysis. Univariate analysis using the selected factors individually as fixed effects and multivariate analysis with appropriate variable selection will be considered, and the hazard ratios and their confidence intervals and p-values will be output from the estimated parameters. Candidate factors shall be as follows.

- Cytogenetic risk group: High Risk 1.
- Components of Frailty adjusted group (Age, ADL, IDAL, CCI) 2.
- Prior antineoplastic therapies\* [Treated, Not treated] 3.
- \*Bortezomib, Carfilzomib, Lenalidomide, Pomalidomide, Elotuzumab, Daratumumab
- Determination of prior treatment efficacy [Clinical relapse, Paraprotein relapse] 4.
- 5. Number of regimens [1, 2, 3 or more)
- ECOG performance status [0, 1, 2, 3, 4] 6.
- LDH 7.
- 8. SEX
- Extramedullary Masses 9.
- Prior hematopoietic stem cell transplantation 10.
- M-protein isotype [IgG  $\kappa \cdot \lambda$ , IgA  $\kappa \cdot \lambda$ , IgD  $\kappa \cdot \lambda$ , IgE  $\kappa \cdot \lambda$ , IgM  $\kappa \cdot \lambda$ , Bence 11. Jones type  $\kappa \cdot \lambda$ , non-secretory type, unknown, others]
- .rum FLC (t
  .<=Max]))
  .5. Renal function Serum FLC (free light chain) (FLC  $\kappa$ , FLC  $\lambda$ ,  $\kappa/\lambda$  ratio [Min<= - <0.26, 0.26=< - <=1.65,

# 7 **SAFETY ANALYSIS**

# subject to the applicable Terms of Use 7.1 Frequency of Treatment-Emergent Adverse Event

# **Overview of Treatment-Emergent Adverse Event** 7.1.1

Analysis Set:

Safety Analysis Set

Analysis Variables:

**TEAE** 

# Category:

Relationship to IRd treatment [Related, Not related] Relationship to study drug [Related, Not related]

Grade [Grade1 – Grade5]

- 1) Frequency count of All TEAEs
- Frequency count of IRd Treatment-related TEAEs 2)
- Frequency count of Study Drug-related TEAEs
  Frequency count of Grade 3 or Higher TEAEs 3)
- 4)
- Frequency count of IRd Treatment-related Grade 3 or Higher TEAEs 5)
- Frequency count of All TEAEs by Grade 6)
- Frequency count of IRd Treatment-related TEAEs by Grade 7)
- Frequency count of Study Drug-related TEAEs by Grade 8)
- Frequency count of TEAEs Resulting in Discontinuation of Treatment 9)
- Frequency count of Serious TEAEs 10)
- Frequency count of Non-serious TEAEs 11)
- Frequency count of TEAEs Resulting in Death 12)

Note for calculation of incidence rate:

· For tabulation by grade

If a patient had two or more adverse events in the same category with different severities, then the event with the maximum severity was used for that patient. The denominator of incidence rate is the number of patients in analysis set.

• Otherwise

If a patient had two or more adverse events in the same category with different severities, then the event with the maximum severity was used for that patient. The denominator of incidence rate is the number of patients in analysis set.

# 7.1.2 **Output of Treatment-Emergent Adverse Event**

Analysis Set:

Safety Analysis Set

Analysis Variables:

**TEAE** 

Category:

Relationship to IRd treatment [Related, Not related]

Relationship to study drug [Related, Not related]

Grade [Grade1 – Grade5]

icable Terms of Use TEAE will be coded using MedDRA and will be summarized by Preferred Term (PT) and System Organ Class (SOC). Analysis output will be sorted SOC alphabetically and PT frequency.

- Frequency count of All TEAEs by SOC and PT 1)
- 2) Frequency count of IRd Treatment-related TEAEs by SOC and PT
- Frequency count of Study Drug-related TEAEs by SOC and PT 3)
- Frequency count of Grade 3 or Higher TEAEs by SOC and PT 4)
- Frequency count of IRd Treatment-related Grade 3 or Higher TEAEs by SOC and PT 5)
- Frequency count of All TEAEs by Grade by SOC and PT 6)
- Frequency count of IRd Treatment-related TEAEs by Grade by SOC and PT 7)
- Frequency count of Study Drug-related TEAEs by Grade by SOC and PT 8)
- Frequency count of TEAEs Resulting in Discontinuation of Treatment by SOC and PT 9)
- Frequency count of Serious TEAEs by SOC and PT 10)
- Frequency count of Non-serious TEAEs by SOC and PT 11)

TEAE that excludes serious TEAE, and the incidence rate exceeds 5 % will be outputted.

Frequency count of TEAEs Resulting in Death by SOC and PT

Note for calculation of incidence rate:

· For tabulation by grade

If a patient had two or more adverse events in the same SOC (or with the same PT) with different severities, then the event with the maximum severity was used for that patient. The denominator of incidence rate is the number of patients in analysis set.

· Otherwise

Patient with two or more AEs in the same SOC (or with the same PT) is counted only once for that SOC (or PT). The denominator of incidence rate is the number of patients in analysis set.

# **Laboratory Results**

Descriptive summary of laboratory data analyzed for safety analysis set.

# **LISTINGS**

Jours or Missing Data

Jours of Missing Data

Jours shall not be imputed unless otherwise noted.

9.3 Criteria for Interim Analysis and Early Discontinuation

All planned analysis will be performed at 12 month after the last patient enrollment.

9.4 Multicenter Studies

Analyses for consideration of medical institution will not be performed.

9.5 Multiple Comparisons/Multiplicity

10 adjustments for multiplicity are p.

1 Consideration

1 Consideration

1 Consideration Multicenter Studies

Analyses for consideration of medical institution will not be performed.

9.5 Multiple Comparisons/Multiplicity

No adjustments for multiplicity are planned.

9.6 Consideration of Subgroups

The subgroups is considered in 6.3.2.

10 REVISION HISTORY

This document is a translation of the 3rd Long.

Acal institution

As/Multiplicity

Aiplicity are planned.

Aion of Subgroups

Are is considered in 6.3.2.

REVISION HISTORY

This document is a translation of the 3rd Japanese version.